CLINICAL TRIAL: NCT07322497
Title: Investigation of the Effects of Video Based Physical Exercise and Physiotherapist Supervised Physical Exercise Before Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison of Video Based Phone App vs. Supervised Preoperative Exercise for ACL Reconstruction
Acronym: ACL-PREHAB-APP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ömer Hekim, Physiotherapist, PhD Candidate, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/23/1304
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament (ACL) Rupture; Anterior Cruciate Ligament (ACL) Reconstruction; Anterior Cruciate Ligament (ACL) Injury
Keywords: Preoperative Rehabilitation; ACL Reconstruciton; Prehabilitation; Mobile Application; Telerehabiltiation
MeSH Terms: conditions — Rupture; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Based App Group (Experimental): Participants will receive a progressive, unsupervised exercise program via a mobile application for 4 weeks prior to surgery. The app provides video guidance, reminders, and compliance tracking.
  Interventions: Behavioral: Mobile App Exercise Program
- Supervised Rehabilitation Group (Active Comparator): Participants will undergo a supervised exercise program with a physiotherapist (3 days/week) for 4 weeks prior to surgery. The protocol is identical to the app group.
  Interventions: Behavioral: Supervised Physiotherapy
- Control Group (No Intervention): Participants will receive standard care and will not receive a specific preoperative exercise prescription.

INTERVENTIONS:
Behavioral: Mobile App Exercise Program — A 4-week progressive home exercise program delivered via a smartphone app. It focuses on range of motion, edema control, strengthening, and balance exercises.
  Arms: Video Based App Group
Behavioral: Supervised Physiotherapy — A 4-week in-clinic exercise program supervised by a physiotherapist, including the same exercises as the app group
  Arms: Supervised Rehabilitation Group

SUMMARY:
The goal of this clinical trial is to learn if using a phone app for exercises is as effective as working with a physical therapist before anterior cruciate ligament knee surgery. It will also check if exercising before surgery helps patients recover better compared to those who do not follow a specific exercise plan. The main questions it aims to answer are:

* Does the phone app help patients improve their knee strength and movement as well as seeing a physical therapist?
* Do patients who exercise before surgery have a better recovery after surgery than those who do not?

Researchers will compare the phone app group to a physical therapist group and a group with no specific exercise plan to see which method works best.

Participants will:

* Follow an exercise plan for 4 weeks before their surgery (either using the app, with a therapist, or no specific plan).
* Visit the clinic for check-ups before starting the exercises, right before the surgery, and 6 months after the surgery.
* Complete simple tests and surveys to measure their knee health.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial designed to investigate the effects of different preoperative rehabilitation methods on patients scheduled for Anterior Cruciate Ligament (ACL) reconstruction.

Participants will be stratified based on their injury type (Isolated ACL injury vs. ACL injury with concomitant meniscus tear) to ensure homogenous distribution. Following stratification, patients will be randomized into three parallel groups using a computer-generated block randomization method (block size of 6).

The study consists of three phases:

1. Pre-operative Intervention (4 Weeks):

   * Video Based Mobile Application Group (Unsupervised): Participants will follow a progressive exercise program via a mobile app. The app provides asynchronous video guidance, reminders, and compliance tracking. The program focuses on range of motion, edema reduction, and muscle strengthening.
   * Supervised Rehabilitation Group: Participants will undergo the exact same exercise protocol under the direct supervision of a physiotherapist (3 sessions/week) in a clinical setting.
   * Control Group: Participants will receive standard care without a specific structured exercise prescription.
2. Surgical Intervention:

   All participants will undergo ACL reconstruction surgery performed by the same surgical team using hamstring autografts.
3. Post-operative Rehabilitation:

Following surgery, ALL patients in all three groups will receive the same standardized, goal based postoperative rehabilitation program. This protocol is based on international criteria and aims to ensure that postoperative care is consistent across all groups, isolating the effect of the preoperative intervention.

Outcomes will be assessed at baseline, preoperatively (after the 4 week program), and 6 months postoperatively. Key assessment methods include:

* Isometric muscle strength testing (Quadriceps and Hamstring) using a hand-held dynamometer.
* Functional performance assessment via Single Leg Hop Tests (limb symmetry index).
* Proprioception evaluation using active joint position sense tests.
* Knee range of motion measurement with a electronic goniometer.
* Patient-reported outcomes using the IKDC 2000 Subjective Knee Evaluation Form.

The primary objective is to determine if the unsupervised digital model is non-inferior to supervised rehabilitation in improving functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosed unilateral Anterior Cruciate Ligament (ACL) rupture
* Patients scheduled for ACL reconstruction surgery.
* Age between 18 and 45 years.
* Patients willing to participate and sign the informed consent form.

Exclusion Criteria:

* Patients with multiple ligament injuries (e.g., combined ACL and PCL/MCL injury).
* Patients with bilateral ACL injuries.
* Presence of accompanying fractures around the knee joint.
* Presence of active infection.
* Patients who refuse surgery or withdraw consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
Isometric Quadriceps Muscle Strength | Baseline, Preoperative (Week 4), and Postoperative (Month 6)
  Muscle strength will be measured using a hand-held dynamometer (Newton). Measurements will be taken at 30 and 70 degrees of knee flexion. The highest value of 3 trials will be recorded.
Isometric Hamstring Muscle Strength | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Muscle strength will be measured using a hand-held dynamometer (Newton) at 35 and 60 degrees of flexion

SECONDARY OUTCOMES:
IKDC 2000 Subjective Knee Evaluation Form | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  A patient-reported outcome measure evaluating knee symptoms and function. Scores range from 0 to 100, with higher scores indicating better function
Knee Range of Motion (ROM) | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Active knee flexion and extension will be measured using a electronic goniometer (degrees)
Single Leg Hop Test (Limb Symmetry Index) | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Participants will hop as far as possible on a single leg. The distance is measured in cm. The Limb Symmetry Index (LSI) will be calculated by comparing the operated leg to the healthy leg.
Star Excursion Balance Test (SEBT) | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Dynamic balance will be assessed by reaching in anterior, posteromedial, and posterolateral directions. Reach distances will be normalized to leg length.
Active Joint Position Sense | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Proprioception will be assessed by the ability to actively reproduce a target angle (15 and 45 degrees) with eyes closed. Absolute angular error will be recorded.
Knee Effusion (Sweep Test) | Baseline, Preoperative (Week 4), and Postoperative (Month 6).
  Joint effusion will be graded on a scale of 0 to 3+ using the Sweep Test technique
Exercise Adherence | Preoperative (Week 4).
  Adherence will be tracked via the mobile app logs (for the app group) and exercise diaries (for the supervised group). It is defined as the percentage of completed prescribed sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No